CLINICAL TRIAL: NCT01891201
Title: Intrapartum Oxytocin Administration Affects Primitive Neonatal Reflexes
Status: Completed | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Miguel Angel Marin Gabriel, MD Pediatrics-Neonatology, Puerta de Hierro University Hospital
Other Study IDs: PI10/00791
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Bonding; Oxytocin; Breastfeeding; Newborn; Perinatal
Keywords: Bonding; Oxytocin; Breastfeeding; Newborn; Delivery
MeSH Terms: conditions — Breast Feeding | interventions — Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Not exposed to oxytocin: Mother-child dyads in which Oxt had not been administered during the birth process
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Comparison of Primitive Newborn Reflexes between those exposed or not to Oxytocin

SUMMARY:
The aim of this study was to assess whether administration of oxytocin intrapartum (Oxt) has any effect on Neonatal Primitive Reflexes (RNP) and if dose dependent. The secondary objective is to assess the effects on exclusive breastfeeding at 3 months

DETAILED DESCRIPTION:
Patients and Methods Prospective case-control study performed in a tertiary hospital. Cases: mother-child dyads in which Oxt had been administered during the birth process (n = 53). Controls: mother-child dyads without Oxt (n = 45). The RNP were recorded with a camcorder in biological nurturing position. An observer blinded to the group and the dose of Oxt codified the RNP (reach/not reached). To assess the type of breastfeeding telephone call was made at 3 months old RN.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton term infant delivered vaginally with Apgar at 5 min> 7;
* Expressed desire to administer during pregnancy breastfeeding;
* Signed informed consent

Exclusion Criteria:

* Preterm neonate;
* Fetal chromosomal or other abnormalities diagnosed in utero to modify their adaptation to extrauterine environment;
* Hospitalization of the mother in ICU;
* Hospitalization in the following 48 hours neonate at birth;
* Wish to artificial feeding before parturition;
* Language difficulties;
* Completion of caesarean delivery

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Maternity ward of a terciary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Expression of Neonatal Primitive Reflexes (RNP) are modified by administration of Oxytocin during delivery. | 72 hours
  Neonatal Primitive Reflexes studied were: 1) Endogenous: hand to mouth, extension / flexion of fingers, mouth open, tongue extrusion, arm circular motion, circular motion of the leg, flex foot / hand, 2) Antigravity: raise the head, 3) Motors: turn your head, nod, plantar pressure, Babinski, and 4) Rhythmic: suction, jaw movement and swallowing.
  An observer, blinded to the study group and the dose administered of Oxytocin, valued recordings, analyzing the state of consciousness at the beginning of the recording as Brazelton scale and form RNP dichotomous coding (achieved / not achieved).

SECONDARY OUTCOMES:
Oxytocin intrapartum may have adverse influence on exclusive breastfeeding at 3 months. | 6 months
  To assess the type of feeding (exclusive breastfeeding versus other) at different time points (discharge, one month and three months) a telephone call was conducted at 3 months old of the newborn.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Marín, MD, Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Madrid, Madrid, Spain

REFERENCES:
- [Background] Carter CS, Williams JR, Witt DM, Insel TR. Oxytocin and social bonding. Ann N Y Acad Sci. 1992 Jun 12;652:204-11. doi: 10.1111/j.1749-6632.1992.tb34356.x. PMID 1626829
- [Background] Carter CS. Developmental consequences of oxytocin. Physiol Behav. 2003 Aug;79(3):383-97. doi: 10.1016/s0031-9384(03)00151-3. PMID 12954433
- [Background] Insel TR, Young LJ. The neurobiology of attachment. Nat Rev Neurosci. 2001 Feb;2(2):129-36. doi: 10.1038/35053579. PMID 11252992
- [Background] Baumgartner T, Heinrichs M, Vonlanthen A, Fischbacher U, Fehr E. Oxytocin shapes the neural circuitry of trust and trust adaptation in humans. Neuron. 2008 May 22;58(4):639-50. doi: 10.1016/j.neuron.2008.04.009. PMID 18498743
- [Background] Ishak WW, Kahloon M, Fakhry H. Oxytocin role in enhancing well-being: a literature review. J Affect Disord. 2011 Apr;130(1-2):1-9. doi: 10.1016/j.jad.2010.06.001. Epub 2010 Jul 2. PMID 20584551
- [Background] Bell AF, White-Traut R, Rankin K. Fetal exposure to synthetic oxytocin and the relationship with prefeeding cues within one hour postbirth. Early Hum Dev. 2013 Mar;89(3):137-43. doi: 10.1016/j.earlhumdev.2012.09.017. Epub 2012 Oct 16. PMID 23084698
- [Background] Malek A, Blann E, Mattison DR. Human placental transport of oxytocin. J Matern Fetal Med. 1996 Sep-Oct;5(5):245-55. doi: 10.1002/(SICI)1520-6661(199609/10)5:53.0.CO;2-H. PMID 8930795
- [Background] Wahl RU. Could oxytocin administration during labor contribute to autism and related behavioral disorders?--A look at the literature. Med Hypotheses. 2004;63(3):456-60. doi: 10.1016/j.mehy.2004.03.008. PMID 15288368
- [Background] Bales KL, Lewis-Reese AD, Pfeifer LA, Kramer KM, Carter CS. Early experience affects the traits of monogamy in a sexually dimorphic manner. Dev Psychobiol. 2007 May;49(4):335-42. doi: 10.1002/dev.20216. PMID 17455224
- [Background] Widstrom AM, Ransjo-Arvidson AB, Christensson K, Matthiesen AS, Winberg J, Uvnas-Moberg K. Gastric suction in healthy newborn infants. Effects on circulation and developing feeding behaviour. Acta Paediatr Scand. 1987 Jul;76(4):566-72. doi: 10.1111/j.1651-2227.1987.tb10522.x. PMID 3630673
- [Background] Righard L, Alade MO. Effect of delivery room routines on success of first breast-feed. Lancet. 1990 Nov 3;336(8723):1105-7. doi: 10.1016/0140-6736(90)92579-7. PMID 1977988
- [Background] Bu'Lock F, Woolridge MW, Baum JD. Development of co-ordination of sucking, swallowing and breathing: ultrasound study of term and preterm infants. Dev Med Child Neurol. 1990 Aug;32(8):669-78. doi: 10.1111/j.1469-8749.1990.tb08427.x. PMID 2210082
- [Background] Olza Fernandez I, Marin Gabriel M, Malalana Martinez A, Fernandez-Canadas Morillo A, Lopez Sanchez F, Costarelli V. Newborn feeding behaviour depressed by intrapartum oxytocin: a pilot study. Acta Paediatr. 2012 Jul;101(7):749-54. doi: 10.1111/j.1651-2227.2012.02668.x. Epub 2012 Apr 4. PMID 22452314
- [Background] Hernandez Aguilar MT, Aguayo Maldonado J; Comite de Lactancia Materna de la Asociacion Espanola de Pediatria. [Breastfeeding. How to promote and support breastfeeding in pediatric practice. Recommendations of the Breastfeeding Committee of the Spanish Association of Pediatrics]. An Pediatr (Barc). 2005 Oct;63(4):340-56. doi: 10.1157/13079817. No abstract available. Spanish. PMID 16219255
- [Background] Torvaldsen S, Roberts CL, Simpson JM, Thompson JF, Ellwood DA. Intrapartum epidural analgesia and breastfeeding: a prospective cohort study. Int Breastfeed J. 2006 Dec 11;1:24. doi: 10.1186/1746-4358-1-24. PMID 17134489
- [Background] Jordan S, Emery S, Watkins A, Evans JD, Storey M, Morgan G. Associations of drugs routinely given in labour with breastfeeding at 48 hours: analysis of the Cardiff Births Survey. BJOG. 2009 Nov;116(12):1622-9; discussion 1630-2. doi: 10.1111/j.1471-0528.2009.02256.x. Epub 2009 Sep 1. PMID 19735379
- [Background] Wiklund I, Norman M, Uvnas-Moberg K, Ransjo-Arvidson AB, Andolf E. Epidural analgesia: breast-feeding success and related factors. Midwifery. 2009 Apr;25(2):e31-8. doi: 10.1016/j.midw.2007.07.005. Epub 2007 Nov 5. PMID 17980469
- [Background] Colson SD, Meek JH, Hawdon JM. Optimal positions for the release of primitive neonatal reflexes stimulating breastfeeding. Early Hum Dev. 2008 Jul;84(7):441-9. doi: 10.1016/j.earlhumdev.2007.12.003. Epub 2008 Feb 19. PMID 18243594
- [Background] Ryden G, Sjoholm I. Half-life of oxytocin in blood of pregnant and non-pregnant women. Acta Endocrinol (Copenh). 1969 Jul;61(3):425-31. No abstract available. PMID 5820054
- [Background] Ermisch A, Barth T, Ruhle HJ, Skopkova J, Hrbas P, Landgraf R. On the blood-brain barrier to peptides: accumulation of labelled vasopressin, DesGlyNH2-vasopressin and oxytocin by brain regions. Endocrinol Exp. 1985 Mar;19(1):29-37. PMID 3872788
- [Background] Ross HE, Young LJ. Oxytocin and the neural mechanisms regulating social cognition and affiliative behavior. Front Neuroendocrinol. 2009 Oct;30(4):534-547. doi: 10.1016/j.yfrne.2009.05.004. Epub 2009 May 28. PMID 19481567
- [Background] Feldman R. Oxytocin and social affiliation in humans. Horm Behav. 2012 Mar;61(3):380-91. doi: 10.1016/j.yhbeh.2012.01.008. Epub 2012 Jan 20. PMID 22285934
- [Background] Febo M, Numan M, Ferris CF. Functional magnetic resonance imaging shows oxytocin activates brain regions associated with mother-pup bonding during suckling. J Neurosci. 2005 Dec 14;25(50):11637-44. doi: 10.1523/JNEUROSCI.3604-05.2005. PMID 16354922
- [Background] Francis DD, Champagne FC, Meaney MJ. Variations in maternal behaviour are associated with differences in oxytocin receptor levels in the rat. J Neuroendocrinol. 2000 Dec;12(12):1145-8. doi: 10.1046/j.1365-2826.2000.00599.x. PMID 11106970
- [Background] Champagne F, Diorio J, Sharma S, Meaney MJ. Naturally occurring variations in maternal behavior in the rat are associated with differences in estrogen-inducible central oxytocin receptors. Proc Natl Acad Sci U S A. 2001 Oct 23;98(22):12736-41. doi: 10.1073/pnas.221224598. Epub 2001 Oct 16. PMID 11606726
- [Background] Winslow JT, Insel TR. The social deficits of the oxytocin knockout mouse. Neuropeptides. 2002 Apr-Jun;36(2-3):221-9. doi: 10.1054/npep.2002.0909. PMID 12359512
- [Background] Klenerova V, Krejci I, Sida P, Hlinak Z, Hynie S. Oxytocin and carbetocin effects on spontaneous behavior of male rats: modulation by oxytocin receptor antagonists. Neuro Endocrinol Lett. 2009;30(3):335-42. PMID 19855356
- [Background] Robinson C, Schumann R, Zhang P, Young RC. Oxytocin-induced desensitization of the oxytocin receptor. Am J Obstet Gynecol. 2003 Feb;188(2):497-502. doi: 10.1067/mob.2003.22. PMID 12592262
- [Background] Phaneuf S, Rodriguez Linares B, TambyRaja RL, MacKenzie IZ, Lopez Bernal A. Loss of myometrial oxytocin receptors during oxytocin-induced and oxytocin-augmented labour. J Reprod Fertil. 2000 Sep;120(1):91-7. doi: 10.1530/jrf.0.1200091. PMID 11006150
- [Background] Gimpl G, Fahrenholz F. The oxytocin receptor system: structure, function, and regulation. Physiol Rev. 2001 Apr;81(2):629-83. doi: 10.1152/physrev.2001.81.2.629. PMID 11274341
- [Background] Phaneuf S, Asboth G, Carrasco MP, Europe-Finner GN, Saji F, Kimura T, Harris A, Lopez Bernal A. The desensitization of oxytocin receptors in human myometrial cells is accompanied by down-regulation of oxytocin receptor messenger RNA. J Endocrinol. 1997 Jul;154(1):7-18. doi: 10.1677/joe.0.1540007. PMID 9246933
- [Background] Olszewski PK, Klockars A, Olszewska AM, Fredriksson R, Schioth HB, Levine AS. Molecular, immunohistochemical, and pharmacological evidence of oxytocin's role as inhibitor of carbohydrate but not fat intake. Endocrinology. 2010 Oct;151(10):4736-44. doi: 10.1210/en.2010-0151. Epub 2010 Aug 4. PMID 20685878
- [Background] Olszewski PK, Klockars A, Schioth HB, Levine AS. Oxytocin as feeding inhibitor: maintaining homeostasis in consummatory behavior. Pharmacol Biochem Behav. 2010 Nov;97(1):47-54. doi: 10.1016/j.pbb.2010.05.026. Epub 2010 Jun 2. PMID 20595062
- [Background] Arletti R, Benelli A, Bertolini A. Oxytocin inhibits food and fluid intake in rats. Physiol Behav. 1990 Dec;48(6):825-30. doi: 10.1016/0031-9384(90)90234-u. PMID 2087513
- [Background] Patient C, Davison JM, Charlton L, Baylis PH, Thornton S. The effect of labour and maternal oxytocin infusion on fetal plasma oxytocin concentration. Br J Obstet Gynaecol. 1999 Dec;106(12):1311-3. doi: 10.1111/j.1471-0528.1999.tb08188.x. PMID 10609728
- [Background] Anagnostakis D, Messaritakis J, Damianos D, Mandyla H. Blood-brain barrier permeability in "healthy" infected and stressed neonates. J Pediatr. 1992 Aug;121(2):291-4. doi: 10.1016/s0022-3476(05)81207-7. PMID 1640301
- [Background] Noseworthy MD, Bray TM. Effect of oxidative stress on brain damage detected by MRI and in vivo 31P-NMR. Free Radic Biol Med. 1998 Apr;24(6):942-51. doi: 10.1016/s0891-5849(97)00383-3. PMID 9607604
- [Background] Jonas W, Johansson LM, Nissen E, Ejdeback M, Ransjo-Arvidson AB, Uvnas-Moberg K. Effects of intrapartum oxytocin administration and epidural analgesia on the concentration of plasma oxytocin and prolactin, in response to suckling during the second day postpartum. Breastfeed Med. 2009 Jun;4(2):71-82. doi: 10.1089/bfm.2008.0002. PMID 19210132
- [Background] Ounsted MK, Hendrick AM, Mutch LM, Calder AA, Good FJ. Induction of labour by different methods in primiparous women. I Some perinatal and postnatal problems. Early Hum Dev. 1978 Sep;2(3):227-39. doi: 10.1016/0378-3782(78)90027-0. PMID 551927
- [Background] Rahm VA, Hallgren A, Hogberg H, Hurtig I, Odlind V. Plasma oxytocin levels in women during labor with or without epidural analgesia: a prospective study. Acta Obstet Gynecol Scand. 2002 Nov;81(11):1033-9. doi: 10.1034/j.1600-0412.2002.811107.x. PMID 12421171
- [Derived] Marin Gabriel MA, Olza Fernandez I, Malalana Martinez AM, Gonzalez Armengod C, Costarelli V, Millan Santos I, Fernandez-Canadas Morillo A, Perez Riveiro P, Lopez Sanchez F, Garcia Murillo L. Intrapartum synthetic oxytocin reduce the expression of primitive reflexes associated with breastfeeding. Breastfeed Med. 2015 May;10(4):209-13. doi: 10.1089/bfm.2014.0156. Epub 2015 Mar 18. PMID 25785487